CLINICAL TRIAL: NCT00816712
Title: A Randomized, Single-Blind, Placebo-Controlled, Single-dose, Parallel Design Study to Evaluate the Effect of Testosterone on Muscle Fractional Synthetic Rate (FSR)
Brief Title: A Study to Evaluate the Effect of Testosterone on Muscle Fractional Synthetic Rate (MK-0000-064)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-064; 2008_604
Record Dates: First submitted 2008-12-31; First posted 2009-01-05 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Muscle Anabolism
Keywords: Males with low-normal serum total testosterone levels.
MeSH Terms: interventions — Injections, Intramuscular

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- A (Active Comparator): Testosterone - 300 mg IM
  Interventions: Drug: Comparator: Testosterone 300 mg, intramuscular injection
- B (Active Comparator): Testosterone - 100 mg IM
  Interventions: Drug: Comparator: Testosterone 100 mg, Intramuscular injection
- C (Placebo Comparator): Placebo - IM
  Interventions: Drug: Comparator: Placebo given by Intramuscular Injection

INTERVENTIONS:
Drug: Comparator: Testosterone 300 mg, intramuscular injection — Day 1 & 7 - Infusion with radioactive tracer (dye), given over 12 hours, followed by two thigh muscle needle biopsies.
  Day 1 & 7 - Testosterone 300 mg, Intramuscular injection.
  Arms: A
Drug: Comparator: Testosterone 100 mg, Intramuscular injection — Day 1 & 7- Infusion with radioactive tracer (dye), given over 12 hours, followed by two thigh muscle needle biopsies.
  Day 1 & 7 - Testosterone 100 mg, Intramuscular injection.
  Arms: B
Drug: Comparator: Placebo given by Intramuscular Injection — Day 1 & 7 - Infusion with radioactive tracer (dye), given over 12 hours, followed by two thigh muscle needle biopsies.
  Day 1 & 7 - Placebo given as intramuscular injection.
  Arms: C

SUMMARY:
This is a study to evaluate the use of fractional synthetic rate as an early biomarker of muscle anabolism (muscle build-up).

ELIGIBILITY:
Inclusion Criteria:

* Subject is weight stable over the past 3 months
* Patient agrees to refrain from consumption of alcohol from 48 hours prior to entering the study
* Subject agrees to follow the study restriction of no caffeine while on study
* Patient agrees to following the meat-free controlled protein weight-maintaining diet
* Patient is willing to avoid strenuous physical activity
* Patient has been a nonsmoker for at least 6 months prior to study start

Exclusion Criteria:

* Subject is currently a regular user of any illicit drugs
* Subject has taken androgenic steroids in the previous 12 months
* Subject has participated in sports events, resistance exercise training or heavy exercise in the previous month
* Subject has prostate cancer
* Subject has a history of cancer except basal-cell tumors
* Subject has been diagnosed with HIV
* Subject has been diagnosed with Hepatitis B or C
* Subject uses certain anti-inflammatory drugs such as ibuprofen, arcoxia or celecoxib
* Subject uses a blood anticoagulant, such as Coumadin (Warfarin) or high doses of aspirin
* Subject is currently taking over the counter supplements such as "muscle builders" or "fat burners"
* Subject has an allergy or hypersensitivity to intramuscular testosterone
* Subject has sciatica
* Subject has donated blood products or has had phlebotomy within 2 months of signing informed consent
* Subject has undergone a surgical procedure within 1 month of signing informed consent
* Subject is currently participating or has participated in a study with an investigational drug or device

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Thigh (vastus lateralis) muscle protein fractional synthetic rate one week after dosing with testosterone. | One week

SECONDARY OUTCOMES:
Variability in the muscle fractional synthetic rate measurements. | One week

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Chen F, Lam R, Shaywitz D, Hendrickson RC, Opiteck GJ, Wishengrad D, Liaw A, Song Q, Stewart AJ, Cummings CE, Beals C, Yarasheski KE, Reicin A, Ruddy M, Hu X, Yates NA, Menetski J, Herman GA. Evaluation of early biomarkers of muscle anabolic response to testosterone. J Cachexia Sarcopenia Muscle. 2011 Mar;2(1):45-56. doi: 10.1007/s13539-011-0021-y. Epub 2011 Feb 26. PMID 21475673